CLINICAL TRIAL: NCT03608150
Title: Luminopia One Amblyopia Vision Improvement Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luminopia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-AM-2
Record Dates: First submitted 2018-07-12; First posted 2018-07-31 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Therapeutic Group (Experimental): Participants assigned to the therapeutic group will be prescribed Luminopia One for 1 hour per day, 6 days per week for 12 weeks.
  Interventions: Device: Luminopia One
- Control Group (Active Comparator): Participants assigned to the control group will wear their current refractive correction full-time for 12 weeks.
  Interventions: Device: Refractive Correction

INTERVENTIONS:
Device: Luminopia One — Luminopia One is a virtual-reality based digital therapeutic that applies therapeutic modifications in real-time to cinematic content to rebalance visual input and treat amblyopia.
  Arms: Therapeutic Group
Device: Refractive Correction — Standard of care refractive correction (ex. spectacles)
  Arms: Control Group

SUMMARY:
The objective of the study is to demonstrate the safety and efficacy of Luminopia One in amblyopia patients with amblyopia associated with anisometropia and/or with mild strabismus.

DETAILED DESCRIPTION:
The proposed study is a multi-center randomized controlled clinical trial which compares the mean change in amblyopic eye Best Corrected Visual Acuity from baseline with Luminopia One ("therapeutic") to refractive correction ("control"). One-hundred and forty participants (n = 140) aged 4-7 years will be enrolled. Participants will be randomized 1:1 to the "therapeutic group ", to use Luminopia One, or the "control group", to undergo continued refractive correction, for 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 7 years at the time of consent.
* Amblyopia associated with anisometropia and/or mild strabismus.
* Current refractive correction worn for at least 16 weeks or until 2 consecutive visual acuity measurements at least 8 weeks apart do not change by more than 1 logMAR lines.
* Amblyopic eye best-corrected visual acuity (BCVA) 20/40 to 20/200 inclusive.
* Fellow eye BCVA 20/32 or better.
* Interocular difference ≥ 3 logMAR lines.
* Heterotropia ≤ 5 prism diopters in current refractive correction at distance measured by SPCT.

Exclusion Criteria:

* Atropine treatment in the past 2 weeks.
* Prior amblyopia treatment (other than refractive correction) for > 12 months in total.
* High myopia, previous intraocular / refractive surgery, severe ocular co-morbidities or development / cognitive delay.
* History of low adherence with amblyopia treatment or light-induced seizures.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Xiao, Study Director — Luminopia
Locations (21):
- United States (21):
  - UCLA Jules Stein Eye Institute, Los Angeles, California
  - Family Focus Eye Care, Gainesville, Florida
  - Eye Physicians of Central Florida, Maitland, Florida
  - Lurie Children's Hospital, Chicago, Illinois
  - IU School of Optometry, Bloomington, Indiana
  - Kids Eye Care of Maryland, Frederick, Maryland
  - Specialized Pediatric Eye Care, Beverly, Massachusetts
  - Children's Eye Care of Michigan, Dearborn, Michigan
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OSU College of Optometry, Columbus, Ohio
  - Pediatric Ophthalmology of Erie, Erie, Pennsylvania
  - Conestoga Eye, Lancaster, Pennsylvania
  - Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Tri-County Eye Physicians, Southampton, Pennsylvania
  - Houston Eye Associates, Houston, Texas
  - Texas Children's Hospital (BCM), Houston, Texas
  - Rocky Mountain Eye Care, Salt Lake City, Utah
  - Virginia Pediatric Eye Center, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapeutic Group | Control Group
Started | 58 | 59
Completed | 47 | 48
Not Completed | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Group | Control Group | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.2 (0.9) | 5.9 (1.1) | 6.0 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 35 | 31 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 6 | 19
  Not Hispanic or Latino | 45 | 53 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 6 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 7 | 11
  White | 50 | 46 | 96
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 117
Prior Amblyopia Treatment [Number; unit: participants] | 48 | 43 | 91

OUTCOME MEASURES:

1. Primary Outcome: Best-Corrected Visual Acuity of Amblyopic Eye
Description: Mean improvement in best-corrected visual acuity of amblyopic eye from baseline after 12 weeks of treatment using electronic ATS-HOTV protocol.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Lines of visual acuity improvement
Arm/Group | Therapeutic Group | Control Group
Number analyzed (Participants) | 47 | 48
Lines of visual acuity improvement | 1.77 (1.56) | 0.85 (1.34)

2. Primary Outcome: Best-Corrected Visual Acuity of Fellow Eye
Description: Mean improvement in best-corrected visual acuity of fellow eye from baseline after 12 weeks of treatment using electronic ATS-HOTV protocol.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Lines of visual acuity improvement
Arm/Group | Therapeutic Group | Control Group
Number analyzed (Participants) | 47 | 48
Lines of visual acuity improvement | 0.30 (0.78) | 0.17 (0.56)

3. Secondary Outcome: Adherence
Description: Mean adherence with the therapeutic in treatment group.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of prescribed therapy
Arm/Group | Therapeutic Group
Number analyzed (Participants) | 56
percentage of prescribed therapy | 85 [48 to 99]

4. Secondary Outcome: Best-Corrected Visual Acuity of Amblyopic Eye
Description: Mean improvement in best-corrected visual acuity of amblyopic eye from baseline after 4 weeks using electronic ATS-HOTV protocol.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Lines of visual acuity improvement
Arm/Group | Therapeutic Group | Control Group
Number analyzed (Participants) | 50 | 49
Lines of visual acuity improvement | 1.06 (1.32) | 0.37 (1.75)

5. Secondary Outcome: Best-Corrected Visual Acuity of Amblyopic Eye
Description: Mean improvement in best-corrected visual acuity of amblyopic eye from baseline after 8 weeks using electronic ATS-HOTV protocol.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Lines of visual acuity improvement
Arm/Group | Therapeutic Group | Control Group
Number analyzed (Participants) | 48 | 44
Lines of visual acuity improvement | 1.48 (1.25) | 0.95 (1.63)

6. Secondary Outcome: Stereoacuity
Description: Mean stereoacuity improvement from baseline after 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Change in log arc seconds
Arm/Group | Therapeutic Group | Control Group
Number analyzed (Participants) | 42 | 46
Change in log arc seconds | 1.0 (5.8) | 0.8 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study at each follow-up phone call or visit.
Description: Serious and Mortality adverse events are reported for all consented individuals. Non-serious adverse events are reported for all participants in the study according to the As Treated Population. i.e. participants actually using the investigational product or the control group product.
Arm/Group | Therapeutic Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 13/51 | 9/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Group (N=51) | Control Group (N=59)
New heterotropia (Eye disorders) | 4 (4) | 4 (4)
Headache (General disorders) | 8 (9) | 1 (1)
Worsening best-corrected visual acuity (Eye disorders) | 2 (2) | 5 (6)

LIMITATIONS AND CAVEATS:
We evaluated the therapeutic alongside continued refractive correction alone over 12 weeks and we did not compare with patching or atropine penalization, so we do not know the relative safety and efficacy of the therapeutic versus patching or atropine, nor the durability of benefit from the therapeutic. The duration of our study was limited to 12 weeks, which may have biased the results toward superiority of one treatment over the other depending on the time course of responses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT03608150/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT03608150/SAP_001.pdf